CLINICAL TRIAL: NCT03003572
Title: Autoreactive Anti-Ro/SSA IgE To Determine Primary SjögRen's Syndrome's Disease Activity
Acronym: I GET DRY
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1608171; ANSM (Other: 2016-A01851-50)
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Sjögren's syndrome; Immunoglobulin E; Anti-Ro/SSA; Autoimmune disease; Biomarker
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with primary Sjögren's syndrome: Blood samples will be collected at inclusion to determine anti-Ro/SSA IgE titers (Enzyme Linked ImmunoSorbent Assay ELISA) in patients with primary Sjögren's syndrome according to the American-European Consensus Criteria.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples will be collected at inclusion to determine anti-Ro/SSA IgE titers (Enzyme Linked ImmunoSorbent Assay ELISA).

SUMMARY:
Primary Sjögren's syndrome (pSS) can affect various organs, sometimes leads to life-threatening conditions and is always responsible for a decreased quality of life. Its evolution is chronic, with flares and relapses, and the need for reliable biomarkers to be carried out routinely is major in patients' follow-up. Because of the existence of autoreactive immunoglobulins E (IgE) in autoimmune diseases, the recently described role for anti-Ro/SSA antibodies in inducing interferon alpha (IFNα) signaling and the specific pharmacologic properties of IgE, anti-Ro/SSA IgE should be an interesting biomarker to determine pSS's activity. The aim of the study is to evaluate whether the proportion of anti-Ro/SSA IgE positive patients is higher in patients with active disease (i.e. Eular Sjögren Syndrome Disease Activity Index≥ 5). All consecutive patients with pSS (new or already known diagnosis) will be included, Anti-Ro/SSA IgE titers will be determined, the disease's features will be collected (including Eular Sjögren Syndrome Disease Activity Index/Eular Sjogren's Syndrome Patient Reported Index).

ELIGIBILITY:
Inclusion Criteria:

* Primary Sjögren's syndrome according to the American-European Consensus Criteria)
* Informed and having signed the study consent form

Exclusion Criteria:

* Secondary Sjögren's syndrome
* Other systemic autoimmune disease (e.g. rheumatoid arthritis, AntiNeutrophil Antibodies (ANCA) -associated vasculitis, mixed connective tissue disease…)
* Incapacity or refusal to sign the informed consent form
* Incapacity or refusal to perform the follow-up examinations required by the study
* Has received abatacept, sifalimumab, rontalizumab, anifrolumab, belimumab, Tumor Necrosis Factor (TNF) antagonists or interferon during the 6 months prior to the inclusion
* Has any current signs or symptoms of active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Sjögren's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of anti-Ro/SSA IgE positive patients | Day 1
  Comparison of proportion of anti-Ro/SSA IgE positive patients between patients with active pSS and patient without active pSS anti-Ro/SSA IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  Active pSS is defined by Eular Sjögren Syndrome Disease Activity Index (ESSDAI) ≥ 5

SECONDARY OUTCOMES:
Correlation between anti-Ro/SSA IgE titers and pSS's activity. | Day 1
  pSS's activity is defined by Eular Sjögren Syndrome Disease Activity Index (ESSDAI).
  Anti-Ro/SSA IgE titers is measured by serial dilutions of the serum. Anti-Ro/SSA IgE titers is the last dilution whose absorbance (in optical density) is higher than positivity threshold.
Correlation between anti-Ro/SSA IgE positive patients and the symptomatology level | Day 1
  Anti-Ro/SSA IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  The symptomatology level is measured by the Score Eular Sjogren's Syndrome Patient Reported Index (ESSPRI).
  If ESSPRI≥5: symptomatology whose intensity felt by the patient is not acceptable.
  If ESSPRI<5: symptomatology whose intensity felt by the patient is acceptable.
Correlation between anti-Ro/SSA IgE positive patients and onset of lymphoma | 5 years
  Anti-Ro/SSA IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  There is a medical monitoring every years by medical record and/or by phone know that a development of lymphoma.
Correlation between anti-Ro/SSA IgE positive patients and interferon alpha signature | Day 1
  Anti-Ro/SSA IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  Interferon alpha signature level is measured by real-time Polymerase Chain Reaction (PCR). They calculate the average of delta cycle threshold in messenger ribonucleic acid (mRNA) of regulate gene by interferon alpha.
Comparison between anti-Ro/SSA IgE positive patients and clinical and biologic characteristics | Day 1
  Anti-Ro/SSA IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  Composite outcome of clinical and biologic characteristics is describe below.
  Clinical characteristics: type of affected organs, lymphoma medical history, allergic disorders, scores Eular Sjögren Syndrome Disease Activity Index (ESSDAI), Eular Sjogren's Syndrome Patient Reported Index (ESSPRI) and analogue visual scale disease patient and doctor, saliva flow and Schirmer test.
  Biologic characteristics: anti-Ro/SSA IgE titers, rheumatoid factor titers and number of totals lymphocytes and T cluster of differentiation 4 (CD4) lymphocytes.
Comparison between anti-La/SSB IgE positive patients and clinical and biologic characteristics | Day 1
  Anti-La/SSB IgE is measured by an indirect quantitative Enzyme Linked ImmunoSorbent Assay (ELISA).
  Composite outcome of clinical and biologic characteristics is describe below.
  Clinical characteristics: type of affected organs, lymphoma medical history, allergic disorders, scores Eular Sjögren Syndrome Disease Activity Index (ESSDAI), Eular Sjogren's Syndrome Patient Reported Index (ESSPRI) and analogue visual scale disease patient and doctor, saliva flow and Schirmer test.
  Biologic characteristics: anti-La/SSB IgE titers, rheumatoid factor titers and number of totals lymphocytes and T CD4 lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal CATHEBRAS, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - CH Pierre Oudot, Bourgoin
  - CHU Estaing - Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble Alpes, Grenoble
  - Hôpital de la Croix Rousse, Lyon
  - CH Lyon Sud, Lyon
  - Hôpital Edouard Herriot - CHU Lyon, Lyon
  - CHU Reims, Reims
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No